CLINICAL TRIAL: NCT04409054
Title: The Guarding Reflex Anal, Study of the Modulation Function of Rectal Distension
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GREEN GRC_01
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Anorectal Disorder
Keywords: Anal Canal; Reflex; Anorectal Manometry; Fecal incontinence; Electromyography
MeSH Terms: conditions — Rectal Diseases; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing the cough and Valsalva protocol: Patients over 18 years old, consulting in neuro urology departement, undergoing ano rectal manometry in order to explore ano rectal disorders
  Interventions: Other: Cough and Valsalva effort

INTERVENTIONS:
Other: Cough and Valsalva effort — Three increasingly cough effort and three Valsalva type effort at four different volumes of rectal distension (empty rectum, volume for a first sensation of filling, volume for desire to defecate and maximal tolerable volume) while recording the external anal sphincter activity

SUMMARY:
The term Guarding Reflex refers to a progressive, involuntary increase in the external urethral sphincter activity during bladder filling.This is a mechanism of continence, preventing from unwanted urine leakage in situation of stress.

Anal continence is essential, and any impairment of this function can have a severe impact on quality of life. Anal continence at rest is mainly insured by the tone of the internal anal sphincter. The external anal sphincter activity during gradually rectal filling is continuous and varies according to the volume of rectal distension.

During an effort, or a cough, the increasing intra-abdominal pressure is transmitted to the rectum. Increased intra-abdominal pressure during an expiratory against resistance effort proportionally increases the response of the external anal sphincter. The reflex contraction of the EAS is an active mechanism under spinal control, and result in a stronger contraction than a voluntary one. This reflex contraction is the equivalent of "Guarding Reflex" and provides part of the continence in situation of stress.

The main purpose of this study is to research a correlation between the ano rectal distension volume and the external anal sphincter response to a stress.

Patient over eighteen years old, consulting for anorectal manometry examination in order to explore anorectal disorders are included.

Age, sex, ano rectal symptoms, treatments, past history, manometrics data, area under the curve for electromyography activity of the EAS and intercostal muscles during cough with a Valsalva effort are recorded. Slope curve representing the EAS response to stress according to the intercostal activity reflecting cough (intensity response curve) effort are calculated.

The protocol consists in distending the rectum at four different volumes. For each volume, the patient is asked to cough three times gradually, and perform a Valsalva effort three times gradually.

Primary outcome is the difference in curve slope (intensity response curves) between empty rectum and maximal tolerable volume at cough Secondary outcomes are the differences in curve slope between each volume of distension at cough, and Valsalva type effort.

DETAILED DESCRIPTION:
The term Guarding Reflex refers to a progressive, involuntary increase in the external urethral sphincter (EUS) activity during bladder filling. Situations increasing intra-abdominal pressure, as cough, or Valsalva effort, increases this EUS activity. This is a mechanism of continence, preventing from unwanted urine leakage in situation of stress.

Anal continence is essential, and any impairment of this function can have a severe impact on quality of life. The anal canal is composed of the internal anal sphincter (IAS) at the top, with smooth musculature and the external anal sphincter (EAS) at the bottom, with striated musculature. The activity of the external anal sphincter is controlled by sympathetic and somatic innervation. Anal continence at rest is mainly insured by the tone of the internal anal sphincter. The external anal sphincter activity during gradually rectal filling is continuous and varies according to the volume of rectal distension.

During an effort, or a cough, the increasing intra-abdominal pressure is transmitted to the rectum. Increased intra-abdominal pressure during an expiratory against resistance effort proportionally increases the response of the external anal sphincter. The reflex contraction of the EAS is an active mechanism under spinal control, and result in a stronger contraction than a voluntary one. This reflex contraction is the equivalent of "Guarding Reflex" and provides part of the continence in situation of stress.

Previous studies focused on the search of segmental or supra segmental control of this reflex. Few studies have examined factors affecting the modulation of the EAS response during stress.

The main purpose of this study is to research a correlation between the ano rectal distension volume and the external anal sphincter response to a stress.

Patient over eighteen years old, consulting for anorectal manometry examination in order to explore anorectal disorders are included.

Age, sex, ano rectal symptoms, treatments, past history, manometrics data, area under the curve for electromyography activity of the EAS and intercostal muscles during cough with a Valsalva effort are recorded. Slope curve representing the EAS response to stress according to the intercostal activity reflecting cough (intensity response curve) effort are calculated.

The protocol consists in distending the rectum at four different volumes : empty rectum, volume for first sensation of filling, volume for desire to defecate and maximal tolerable volume. For each volume, the patient is asked to cough three times gradually, and perform a Valsalva effort three times gradually.

Primary outcome is the difference in curve slope (intensity response curves) between empty rectum and maximal tolerable volume at cough

Secondary outcomes are the differences in curve slope between each volume of distension at cough, and the differences in curve slope between each volume of distension at Valsalva type effort.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Ano rectal disorders

Exclusion Criteria:

* Inability to understand simple orders
* Anal hypotonia
* Peripheral neurological disorder
* Anal incontinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over eighteen years old consulting in the neuro urology departement for ano rectal disorders, undergoing ano rectal manometry examination
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in curve slope between empty rectum and maximal tolerable volume at cough | 1 day
  The area under the curve of EAS response to stress is recorded three times (at each cough effort) for each volume of distension. Curve representing the intensity response is build for each volume of rectal distension. Then, the curve slopes are compared.

SECONDARY OUTCOMES:
Difference in curve slope between each volume of distension at cough | 1 day
  The area under the curve of EAS response to stress is recorded three times (at each cough effort) for each volume of distension. Curve representing the intensity response is build for each volume of rectal distension. Then, the curve slopes are compared.
Difference in curve slope between each volume of distension at Valsalva type effort. | 1 day
  The area under the curve of EAS response to stress is recorded three times (at each Valsalva type effort) for each volume of distension. Curve representing the intensity response is build for each volume of rectal distension. Then, the curve slopes are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP,Hôpital Tenon, Paris, France
Locations (1):
- Department of neuro-urology, hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided